CLINICAL TRIAL: NCT04643184
Title: Clinical Trial on Follow-up Strategies for Fragile Patients With Decompensated Heart Failure
Brief Title: Follow-up Strategies for Fragile Patients With Decompensated Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment rate
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5452
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; With Decompensation; Fragility
MeSH Terms: conditions — Heart Failure | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Co-management program (cardiological-geriatric) to carry out during hospitalization a comprehensive evaluation that allows to know the medical and socio-environmental needs of the patients to plan the required care at home and achieve an effective transition.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Management Program (Experimental): Comanagement program (cardiological-geriatric) to carry out during hospitalization a comprehensive evaluation that allows to know the medical and socio-environmental needs of the patients to plan the required care at home and achieve an effective transition.
  Interventions: Other: Management Program
- Usual Care (No Intervention): Usual care during hospitalizacion and discharge.

INTERVENTIONS:
Other: Management Program — Joint management between the geriatric and cardiology team of the geriatric syndromes and heart failure. Education of the patient and their caregiver, preparing them for the transition of care.
  Arms: Management Program

SUMMARY:
Randomized controlled clinical trial with intervention branch (management program cardiological-geriatric) and control branch (usual care) for fragile patients with decompensated heart failure.

DETAILED DESCRIPTION:
Randomized controlled clinical trial with intervention branch (management program cardiological-geriatric) and control branch (usual care) for fragile patients with decompensated heart failure. Follow-up period 1 month.

This protocol aims through a multidisciplinary vision, to carry out during hospitalization a comprehensive geriatric evaluation that allows to know the medical and socio-environmental needs of the patient to plan the required care at home and achieve an effective transition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. Decompensated heart failure
3. FRAIL scale equal to 3 or more points
4. Permanent residence in the Metropolitan Area of Buenos Aires

Exclusion Criteria:

1. Refusal to participate in the study
2. Terminal oncology or cardiological disease
3. Reversible or treatable etiology heart failure (e.g. Takotsubo, acute cardiomyocarditis)
4. Patients followed by geriatrics prior to admission
5. Simultaneous participation in another research protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Hospital admission | 30 days
  Number of hospital admission for any cause within 30 days

SECONDARY OUTCOMES:
Mortality | 30 days
  Number of deaths from any cause within 30 days

OTHER OUTCOMES:
Prevalence of fragility | Admission
  The proportion of patients with a FRAIL scale equal to 3 or more points of the total number of patients hospitalized for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: César Belziti, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Rodrigo Aguirre, Buenos Aires, C.a.b.a, Argentina

IPD SHARING:
Plan to Share IPD: No